CLINICAL TRIAL: NCT01470729
Title: Identification of Biomarkers in Patients With Autosomal Dominant Cerebellar Ataxia
Brief Title: Biomarkers in Autosomal Dominant Cerebellar Ataxia
Acronym: BIOSCA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P100125
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2014-06

CONDITIONS: Spinocerebellar Ataxia Type 1; Spinocerebellar Ataxia Type 2; Spinocerebellar Ataxia, Autosomal Recessive 3; Episodic Ataxia, Type 7
Keywords: Spinocerebellar ataxia, energy metabolism, NMR spectroscopy
MeSH Terms: conditions — Spinocerebellar Ataxias; Spinocerebellar ataxia, autosomal recessive 3; Episodic Ataxia, Type 7 | interventions — Metabolic Networks and Pathways

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Spinocerebellar Ataxia type 1 (SCA1): Spinocerebellar Ataxia type 1 (SCA1)
  Interventions: Other: metabolic and imaging biomarkers in SCA1,2,3 and 7 patients
- Spinocerebellar Ataxia type 2 (SCA2): Spinocerebellar Ataxia type 2 (SCA2)
  Interventions: Other: metabolic and imaging biomarkers in SCA1,2,3 and 7 patients
- Spinocerebellar Ataxia type 3 (SCA3): Spinocerebellar Ataxia type 3 (SCA3)
  Interventions: Other: metabolic and imaging biomarkers in SCA1,2,3 and 7 patients
- Spinocerebellar Ataxia type 7 (SCA7): Spinocerebellar Ataxia type 7 (SCA7)
  Interventions: Other: metabolic and imaging biomarkers in SCA1,2,3 and 7 patients

INTERVENTIONS:
Other: metabolic and imaging biomarkers in SCA1,2,3 and 7 patients — MRI, a bone mineral density and a resting metabolic rate assessments, as well as donating fasted blood samples

SUMMARY:
Autosomal dominant cerebellar ataxias (ADCA) are a group of neurodegenerative disorders that are clinically and genetically various. BIOSCA study aims to identify markers of the metabolism (energy production inside the cells) in the blood and the brain of ADCA 1,2,3 and 7 patients and control subjects, in the perspective of future therapeutic trials.

DETAILED DESCRIPTION:
Rational. Autosomal dominant cerebellar ataxias (ADCA) are a clinically heterogeneous group of neurodegenerative disorders caused by unstable CAG repeat expansions encoding polyglutamine tracts. ADCA have a wide range of neurological symptoms including ataxia of gait, stance, and limbs, cerebellar dysarthria, oculomotor disturbances of cerebellar and supranuclear genesis, retinopathy, optic atrophy, spasticity, extra-pyramidal movement disorders, peripheral neuropathy, sphincter disturbances, cognitive impairment, and epilepsy. Corresponding to neuropathological findings in hereditary ataxia, there are three fundamental patterns of degeneration on MRI: spinal atrophy, olivopontocerebellar atrophy, and cortical cerebellar atrophy. We previously showed an hypercatabolism in premanifest and early stage Huntington's disease (HD), along with a systemic metabolic defect: progressive decrease of the plasmatic branched-chain amino acids (BCAA) - correlated with low serum IGF1 (insulin-like growth factor 1) - and muscle energy metabolism abnormalities measured by 31P-NMR spectroscopy. We also observed a weight loss in SCA1, 3 and mostly SCA7 patients. In addition, we underlined in a preliminary study a significant decrease of the BCAA in SCA1,2,3 and 7 patients, suggesting that an energy deficit would also be implied in SCA pathogenesis. Transcriptional interferences are likely a part of SCA physiopathology, as shown in the retinal cells of a SCA7 mouse model, or as we detected over the cerebellum growth of these mice. The hallmark of the gene expression studies in SCA1 and SCA7 mice points out the implication of IGF1 pathway and IGF1 receptor. As in HD, these transcriptional disorders might witness the metabolic defects above-mentioned.

Study objectives. The primary aim of the study is to provide metabolic and imaging biomarkers in SCA1,2,3 and 7 patients and controls in the perspective of future therapeutic trials.

The secondary aims are to determine (i) an systemic energy profile in SCA1,2,3 and 7 patients with the confirmation of an hypercatabolic status, (ii) a brain energy profile in SCA1,2,3 and 7 patients measured by in vivo 31P-NMR spectroscopy.

Study population. BIOSCA will recruit 120 participants in the Pitie Salpetriere University Hospital located in Paris, France. The target cohort will be 80 patients - divided into 4 groups of 20 participants of each mutation - and 40 controls.

Study design. All patients (SCA1,2,3,7) will be assessed at baseline (visit 1), 1 year (visit 2) and 2 years (visit 3). At visit 1 and 3, subjects will undergo clinical, MRI, a bone mineral density and a resting metabolic rate assessments, as well as donating fasted blood samples. Each visit will last approximately 6 hours. At visit 2, they will have only a clinical assessment along with a fasted blood sample. Control subjects will be seen only at visit 1 and 3 with the same assessments as the patients.

Study period. BIOSCA is a prospective study for which each participant is enrolled for 24 months. The study duration is 36 months. The start date is November 2011.

Funding. BIOSCA is funded by a national funding hospital program in clinical research (PHRC) from APHP institution.

ELIGIBILITY:
Inclusion criteria :

* More than 18 years of age
* Ability to tolerate MRI
* Positive genetic test to SCA1, 2, 3 or 7
* Coverage by social insurance
* Written informed consent must be obtained from the subject

Exclusion criteria :

* Less than 18 years of age
* Concomitant significant neurological disorder
* Unsuitability for MRI, e.g. claustrophobia, metal implants
* History of significant head injury
* Unability to receive an informed explanation about the protocol
* Unability to complete the protocol
* Non coverage by social insurance
* No written informed consent obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Spinocerebellar Ataxia Type 1 (SCA1) Spinocerebellar Ataxia Type 2 (SCA2) Spinocerebellar Ataxia Type 3 (SCA3) Spinocerebellar Ataxia Type 7 (SCA7)
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
metabolic biomarkers of SCA | 12 months or 24 months

SECONDARY OUTCOMES:
imaging biomarkers of SCA | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra DURR, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié Salpêtrière, Paris, France

REFERENCES:
- [Result] Adanyeguh IM, Henry PG, Nguyen TM, Rinaldi D, Jauffret C, Valabregue R, Emir UE, Deelchand DK, Brice A, Eberly LE, Oz G, Durr A, Mochel F. In vivo neurometabolic profiling in patients with spinocerebellar ataxia types 1, 2, 3, and 7. Mov Disord. 2015 Apr 15;30(5):662-70. doi: 10.1002/mds.26181. Epub 2015 Mar 15. PMID 25773989
- [Result] Adanyeguh IM, Perlbarg V, Henry PG, Rinaldi D, Petit E, Valabregue R, Brice A, Durr A, Mochel F. Autosomal dominant cerebellar ataxias: Imaging biomarkers with high effect sizes. Neuroimage Clin. 2018 Jun 14;19:858-867. doi: 10.1016/j.nicl.2018.06.011. eCollection 2018. PMID 29922574
- [Result] Garali I, Adanyeguh IM, Ichou F, Perlbarg V, Seyer A, Colsch B, Moszer I, Guillemot V, Durr A, Mochel F, Tenenhaus A. A strategy for multimodal data integration: application to biomarkers identification in spinocerebellar ataxia. Brief Bioinform. 2018 Nov 27;19(6):1356-1369. doi: 10.1093/bib/bbx060. PMID 29106465
- [Derived] Faber J, Schaprian T, Berkan K, Reetz K, Franca MC Jr, de Rezende TJR, Hong J, Liao W, van de Warrenburg B, van Gaalen J, Durr A, Mochel F, Giunti P, Garcia-Moreno H, Schoels L, Hengel H, Synofzik M, Bender B, Oz G, Joers J, de Vries JJ, Kang JS, Timmann-Braun D, Jacobi H, Infante J, Joules R, Romanzetti S, Diedrichsen J, Schmid M, Wolz R, Klockgether T. Regional Brain and Spinal Cord Volume Loss in Spinocerebellar Ataxia Type 3. Mov Disord. 2021 Oct;36(10):2273-2281. doi: 10.1002/mds.28610. Epub 2021 May 5. PMID 33951232
- [Derived] Coarelli G, Darios F, Petit E, Dorgham K, Adanyeguh I, Petit E, Brice A, Mochel F, Durr A. Plasma neurofilament light chain predicts cerebellar atrophy and clinical progression in spinocerebellar ataxia. Neurobiol Dis. 2021 Jun;153:105311. doi: 10.1016/j.nbd.2021.105311. Epub 2021 Feb 23. PMID 33636389